CLINICAL TRIAL: NCT00365937
Title: Immunization of Disease-Free Melanoma Patients With Different HLA-A2 Peptides
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: New regulatories of the peptides by the pharmaceutical company (the seller)
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Immutep S.A.S. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUC 05-003
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Melanoma
Keywords: immunotherapy; adjuvants; IMP321; Montanide ISA51 VG; tumor-specific peptides
MeSH Terms: conditions — Melanoma | interventions — Adjuvants, Immunologic; montanide ISA 51; soluble LAG-3 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): The eight HLA-A2 peptides
  Interventions: Biological: Immunological peptides and immunological adjuvants; Biological: HLA-A2 peptides
- Group B (Experimental): The eight HLA-A2 peptides + immunological adjuvant Montanide ISA51
  Interventions: Biological: Immunological peptides and immunological adjuvants; Biological: HLA-A2 peptides; Biological: Montanide ISA51
- Group C (Experimental): the eight peptides HLA-A2 + IMP321
  Interventions: Biological: Immunological peptides and immunological adjuvants; Biological: HLA-A2 peptides; Biological: IMP321
- Group D (Experimental): The eight HLA-A2 peptides + the 2 immunological adjuvants (Montanides ISA 51 and IMP321)
  Interventions: Biological: Immunological peptides and immunological adjuvants; Biological: HLA-A2 peptides; Biological: Montanide ISA51; Biological: IMP321

INTERVENTIONS:
Biological: Immunological peptides and immunological adjuvants
Biological: HLA-A2 peptides — Tyrosinase.A2: lyophilized powder, 326 mcg, 5 injections every 3 weeks MAGE-C2.A2: lyophilized powder, 320 mcg, 5 injections every 3 weeks NY-ESO-1b.A2: lyophilized powder, 290 mcg, 5 injections every 3 weeks MAGE-4.A2: lyophilized powder, 299 mcg, 5 injections every 3 weeks MAGE-3.A2: lyophilized powder, 300 mcg, 5 injections every 3 weeks MAGE-1.A2: lyophilized powder, 298 mcg, 5 injections every 3 weeks NA17.A2 (GnTV): lyophilized powder, 300 mcg, 5 injections every 3 weeks MAGE-10.A2: lyophilized powder, 309 mcg, 5 injections every 3 weeks
Biological: Montanide ISA51 — Oil emulsion (W/O: droplet test S57 IN 001), conductivity less than 10mcs.cm-1, viscosity: 1500 mPas (brookfield DVI - spindle 2- Speed 30). For human applications. Injected 5 times every 3 weeks.
  Arms: Group B; Group D
Biological: IMP321 — Official name of the LAG-3 molecule is CD223. Chemical structure: hLAG-3Ig is a soluble human recombinant LAG-3 protein comprising the extra-cellular Ig-like domains.
  The IMP321 drug product is composed of a soluble recombinant protein at a 1.18 mg/ml concentration, in PBS (Na2HPO4 2H2O 8.1mM, KH2PO4 1.47mM, NaCl 137mM, KCl 2.68mM, PH 7.2). Batch number: S017/LC1/041011.IMP321 will be provided in 250mcl aliquots in brosilicate siliconized vials.
  Arms: Group C; Group D

SUMMARY:
Open-label single center study. Patients will be divided in four groups of 7. Group 1: 8 melanoma-specific peptides in saline; Group 2: same mix of peptides + Montanide ISA51; Group 3: same mix of peptides + IMP321 500 µg; Group 4: same mix of peptides + IMP321 500 µg + Montanide ISA51. These vaccines will be administered every 3 weeks on 5 occasions by intradermal and superficial subcutaneous injections.

DETAILED DESCRIPTION:
Open-label single center study. Patients will be divided in four groups of 7. The patients will be entered sequentially at the time they present in clinic, and randomized in one of the four groups.

The first group of patients will receive a dose of 300 µg of each of the MAGE-1.A2, MAGE-3.A2, MAGE-4.A2, MAGE-10.A2, MAGE-C2.A2, NA17.A2, Tyrosinase.A2 and NY-ESO-1.A2 peptides without adjuvant. The peptides will be mixed together and administered by intradermal and superficial subcutaneous injections at two sites every three weeks on 5 occasions (3 months).

The second group of patients will receive on 5 occasions a vaccine containing the same 8 peptides mixed together but emulsified in 1 ml of Montanide ISA51. This vaccine will be also administered by intradermal and subcutaneous injections every three weeks.

The third cohort of patients will receive at 3 weeks-interval on 5 occasions the mix of 8 peptides and 500 µg of IMP321. These two injections will be done at the same site, first adjuvant IMP321 then the peptides.

The last seven patients will receive as vaccine the same mix of peptides emulsified with Montanide ISA 51 VG and IMP321 injected with the same procedure as cohort 3. These vaccines will be administrated every 3 weeks on 5 occasions by intradermal and superficial subcutaneous injections.

Blood samples will be obtained from a buffy-coat at weeks 1 and 16. PBL collected at baseline (day 1) and at week 16 will be tested to determine whether a specific CTL response, defined as a 10-times or more increase in CTL frequency, occurred.

For the patients with an anti-vaccine lymphocyte response, 100 ml of blood will be collected every three months in order to monitor their immune response. If a decrease in CTL frequency by a factor 10 is observed, the patients will be revaccinated three times at three weeks interval with the peptide(s) against which he developed an immune response mixed with the adjuvant he already received.

The disease status will be assessed at study entry and thereafter every 3 months during one year. At any time, relapse will result in withdrawal of the patient from the trial.

ELIGIBILITY:
Inclusion Criteria:

Histologically proven cutaneous melanoma.

Patient's melanoma must be in one of the following AJCC stages :

only primary tumor : T3b-T4, N0, M0. regional lymph node metastasis and/or in-transit metastasis, no distant metastasis (any T, N1-N3, M0) that has been removed.

Any distant metastasis that has been removed (M1) HLA-A2 positive. Patients with previous regional metastatic disease must have one of their resected lesions analyzed by RT-PCR to determine expression of genes MAGE-1, MAGE-3, MAGE-4, MAGE-10, MAGE-C2, NA17, Tyrosinase or NY-ESO-1. However, expression of these genes by the tumor is not required to enter the study.

Absence of detectable melanoma lesions. WHO/ECOG performance status of 1 or less (Karnofsky scale ≥ 70%).

The following laboratory results:

Hemoglobin ≥ 10 g/dl; Neutrophils ≥ 1,500/µl; Lymphocytes ≥ 700/µl; Platelets ≥ 100,000/µl; Serum creatinin ≤ 2.0 mg/dl; Serum bilirubin ≤ 2.0 mg/dl; LDH within normal institutional limits.

Age > 18 years. Able to give written informed consent.

Exclusion Criteria:

Clinically significant heart disease (NYHA Class III or IV). Other serious illnesses, e.g. serious infections requiring antibiotics, bleeding disorders, a second active malignancy, except basal cell carcinoma or in situ carcinoma of the uterine cervix.

Active immunodeficiency disease or autoimmune disease. Positive serology for HIV (human immunodeficiency virus) or HCV (hepatitis C virus). Serum hepatitis B antigen (HBsAg) must be negative.

More than one line of previous chemotherapy, or immunotherapy for the melanoma. Previous vaccination with one of the antigen present in the vaccine. Treatment with steroids or major immunosuppressive drugs within 4 weeks before study entry. Topical or inhalational steroids are permitted.

Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.

Pregnancy or lactation. Women of childbearing potential not using a medically acceptable means of contraception.

Psychiatric or addictive disorders that may compromise the ability to give informed consent.

Lack of availability of the patient for immunological and clinical follow-up assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2013-12-13 (Actual); Study Completion 2013-12-13 (Actual)

PRIMARY OUTCOMES:
Primary: Determination of the cytolytic T lymphocyte response in the different arms.; Toxicity of the combination peptide and immunological adjuvants

SECONDARY OUTCOMES:
Secondary: Disease-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Baurain, M.D, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium